CLINICAL TRIAL: NCT00096915
Title: A Multicenter, Single-Arm Study Evaluating Once Monthly Darbepoetin Alfa Dosing in Subjects With Chronic Kidney Disease (CKD) Receiving Dialysis
Brief Title: Study Evaluating Darbepoetin Alfa in Subjects With Chronic Kidney Disease (CKD) Receiving Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20040202
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Last update posted 2009-05-22 (Estimated); Status verified 2009-05

CONDITIONS: Kidney Disease; Chronic Kidney Disease
Keywords: chronic kidney disease, CKD; renal failure; anemia; hemodialysis; peritoneal dialysis; Aranesp®, Darbepoetin Alfa
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic; Renal Insufficiency; Anemia | interventions — Darbepoetin alfa

ARMS (1):
- darbepoetin alfa (Experimental)
  Interventions: Drug: Darbepoetin Alfa

INTERVENTIONS:
Drug: Darbepoetin Alfa — QM administration for 32 weeks, allowable doses:
  15, 20, 30, 40, 50, 60, 80, 100, 150, 200, 300, 400, 500, 600 and 800 mcg

SUMMARY:
The proposed study is designed to test a novel dosing paradigm that would facilitate the treatment of anemia in CKD patients on dialysis. Anemic patients on hemo and peritoneal dialysis who have achieved and maintained target hemoglobin (Hb) on every other week (Q2W) dosing of darbepoetin alfa will have the dosing interval extended to once monthly (QM) dosing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic kidney disease (CKD) and receiving dialysis for > 3 months before enrollment
* Clinically stable, in the judgment of the investigator
* Mean Hb > 11.0 g/dL (110 g/L) to < 13.0 g/dL (130 g/L)
* Transferrin saturation (Tsat) > 19.5%
* Serum vitamin B12 and folate levels above the lower limit of the normal range
* Receiving stable Q2W IV or SC doses of Aranesp® (darbepoetin alfa). A stable dose is defined as less than or equal to 25% change in dose over the 6-week period immediately prior to enrollment and with no missed doses in this period

Exclusion Criteria:

* Scheduled to receive a kidney transplant
* Diastolic blood pressure greater than 110 mm Hg or systolic BP greater than 180 mm Hg during screening
* Acute myocardial ischemia
* Hospitalization for congestive heart failure, myocardial infarction, deep vein thrombosis, stroke or transient ischemic attack within 12 weeks before enrollment
* Parathyroid hormone (PTH) level greater than 1500 pg/mL (158.0 pmol/L)
* Major surgery within 12 weeks before enrollment (excluding vascular access surgery)
* Currently receiving antibiotic therapy for systemic infection
* Known positive HIV antibody or positive hepatitis B surface antigen
* Clinical evidence of current malignancy and/or receiving systemic chemotherapy/radiotherapy with the exception of basal cell or squamous cell carcinoma of the skin and cervical intraepithelial neoplasia
* Red blood cell (RBC) transfusions within 8 weeks before enrollment
* Androgen therapy within 8 weeks before enrollment - Systemic hematologic disease (e.g., sickle cell anemia, myelodysplastic syndromes, hematologic malignancy, myeloma, hemolytic anemia)
* Any disorder that may impact (in the judgment of the investigator) the ability to give informed consent for participation in this study
* Pregnant or breast-feeding women
* All subjects must practice adequate contraception (in the judgment of the investigator) throughout this trial
* Treatment with an investigational agent or device within 30 days before enrollment or scheduled to receive an investigational agent other than those specified by this protocol during the course of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2004-10; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects on QM darbepoetin alfa dosing maintained with a mean Hb greater than or equal to 11.0 g/dL and less than or equal to 13.0 g/dL during the evaluation phase | entire study

SECONDARY OUTCOMES:
Hb values over the duration of the study | entire study
Darbepoetin alfa doses over the duration of the study | entire study
Frequency and relationship to treatment for adverse events and changes in laboratory parameters and blood pressure | entire study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_33_NESP_20040202.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/